CLINICAL TRIAL: NCT01358331
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Efficacy of MK-8353 (Formerly SCH 900353) in Subjects With Advanced Solid Tumors (Protocol No. 001 (Formerly P06203))
Brief Title: A Study of the Safety, Tolerability, and Efficacy of MK-8353 in Participants With Advanced Solid Tumors (MK-8353-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P06203; 2012-002696-33 (EudraCT Number); MK-8353-001 (Other: Merck)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms | interventions — MK-8353

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK-8353 100 mg twice daily (BID) (Experimental): 100 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353
- MK-8353 200 mg BID (Experimental): 200 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353
- MK-6353 300 mg BID (Experimental): 300 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353
- MK-8353 350 mg BID (Experimental): 350 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353
- MK-8353 400 mg BID (Experimental): 400 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353
- MK-8353 800 mg BID (Experimental): 800 mg capsules administered orally twice daily for 28 days for each cycle
  Interventions: Drug: MK-8353

INTERVENTIONS:
Drug: MK-8353 — Administered orally twice daily for 28 days for each cycle

SUMMARY:
This study of the safety, tolerability, and efficacy of MK-8353 (formerly SCH 900353) given as single agent oral therapy for participants with advanced solid tumors will be done into two parts. In Part 1a, there will be a dose escalation to find the preliminary maximum tolerated dose (MTD), and in Part 1b, dose confirmation to find out the recommended Phase 2 dose (RPTD) that will be used in Part 2 of the study. In Part 2 of the study, participants with certain types of metastatic melanoma or metastatic colorectal cancer will be treated to see if MK-8353 is effective as single agent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically/histologically confirmed solid tumor (metastatic or locally advanced disease) that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
* Participants of childbearing potential must have negative pregnancy test; females and males must agree to use effective contraception during the course of the trial and for 90 days after stopping study drug.
* For Part 1b and Part 2, participant with metastatic melanoma or metastatic colorectal cancer with at least one measurable lesion
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with a life expectancy of ≥3 months.
* Adequate organ function.

Exclusion Criteria:

* Unstable or progressing central nervous system (CNS) metastasis unless asymptomatic for 3 months, with no need for steroids or antiseizure medications.
* Active gastrointestinal disease or a disorder or a history of surgery that significantly alters gastrointestinal motility or absorption.
* Has not recovered from previous therapy and had any chemotherapy, biologic, or hormonal therapy within 4 weeks of study enrollment.
* Radiation therapy (except palliative radiation to bone lesions) within 4 weeks of study enrollment.
* More than 3 prior regimens of chemotherapy, biologic therapy, hormonal therapy, or investigational drugs not including adjuvant or neoadjuvant treatments.
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic diseases.
* Mean QTcF interval (interval on the electrocardiogram corrected for heart rate using Fridericia's correction) > 450 msec at baseline.
* Known Human Immunodeficiency Virus (HIV) infection, hepatitis infection, or tuberculosis infection.
* Current participation in any other interventional clinical study.
* History of significant eye disease, including glaucoma, retinopathy, or retinal vein occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2014-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharpe & Dohme Corp.

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Moschos SJ, Sullivan RJ, Hwu WJ, Ramanathan RK, Adjei AA, Fong PC, Shapira-Frommer R, Tawbi HA, Rubino J, Rush TS 3rd, Zhang D, Miselis NR, Samatar AA, Chun P, Rubin EH, Schiller J, Long BJ, Dayananth P, Carr D, Kirschmeier P, Bishop WR, Deng Y, Cooper A, Shipps GW, Moreno BH, Robert L, Ribas A, Flaherty KT. Development of MK-8353, an orally administered ERK1/2 inhibitor, in patients with advanced solid tumors. JCI Insight. 2018 Feb 22;3(4):e92352. doi: 10.1172/jci.insight.92352. eCollection 2018 Feb 22. PMID 29467321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 participants were enrolled, received at least 1 dose of MK-8353 and were included in the analysis.
Groups:
- MK-8353 100 mg Twice Daily (BID): Participants received 100 mg twice daily for 28 days during each cycle
- MK-8353 200 mg BID: Participants received 200 mg twice daily for 28 days during each cycle
- MK-8353 300 mg BID: Participants received 300 mg twice daily for 28 days during each cycle
- MK-8353 350 mg BID: Participants received 350 mg twice daily for 28 days during each cycle
- MK-8353 400 mg BID: Participants received 400 mg twice daily for 28 days during each cycle
- MK-8353 800 mg BID: Participants received 800 mg twice daily for 28 days during each cycle
Period: Overall Study
Arm/Group | MK-8353 100 mg Twice Daily (BID) | MK-8353 200 mg BID | MK-8353 300 mg BID | MK-8353 350 mg BID | MK-8353 400 mg BID | MK-8353 800 mg BID
Started | 2 | 3 | 4 | 3 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 4 | 3 | 7 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Adverse Events | 1 | 1 | 1 | 0 | 1 | 5
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participants did not wish to continue | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progress of disease under investigation | 1 | 2 | 3 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Any participant who received at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8353 100 mg Twice Daily (BID) | MK-8353 200 mg BID | MK-8353 300 mg BID | MK-8353 350 mg BID | MK-8353 400 mg BID | MK-8353 800 mg BID | Total
Number analyzed (Participants) | 2 | 3 | 4 | 3 | 7 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (5.7) | 49.3 (11.4) | 62.5 (8.4) | 64.3 (9.0) | 59.3 (9.3) | 59.8 (9.0) | 59.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 3 | 2 | 9
  Male | 1 | 2 | 3 | 2 | 4 | 4 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 1 | 4 | 3 | 7 | 5 | 22
  Race Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was derived from the toxicities observed during the first cycle (28 days) for each dose level. DLT is defined as any hematologic or non-hematologic toxicity ≥Grade 3 as pre-specified per protocol, or drug-related toxicity, regardless of Common Terminology Criteria for Adverse Events (CTCAE) grade that causes >20% of the intended total number of doses in Cycle 1 to be missed.
Time Frame: Cycles of 28 days, up to approximately 9 months treatment and a 30-day follow-up period for a total time of up to approximately 10 months
Population: Analysis population includes all participants who received at least one dose of MK-8353 and completed Cycle 1 of Part 1 or discontinued due to toxicity. Participants who discontinued treatment due to reasons other than toxicity were not included.
Measure: Number; unit: Participants
Arm/Group | MK-8353 100 mg Twice Daily (BID) | MK-8353 200 mg BID | MK-8353 300 mg BID | MK-8353 350 mg BID | MK-8353 400 mg BID | MK-8353 800 mg BID
Number analyzed (Participants) | 2 | 3 | 4 | 3 | 6 | 2
Participants
  Grade 3 Maculopapular Rash | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Diarrhea | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 fatigue | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 nausea/vomiting/diarrhea | 0 | 0 | 0 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Overall Response Rate
Description: Overall Response rate is defined as the number of participants who had a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Baseline, and every 8 weeks until disease progression or discontinuation from study up to approximately 10 months
Population: The analysis population is defined as all participants who received at least 1 dose of MK-8353 and had at least 1 post-baseline efficacy assessment. Participants who received at least one dose but had no post-baseline assessment were counted as "not evaluable" and were not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | MK-8353 100 mg Twice Daily (BID) | MK-8353 200 mg BID | MK-8353 300 mg BID | MK-8353 350 mg BID | MK-8353 400 mg BID | MK-8353 800 mg BID
Number analyzed (Participants) | 2 | 3 | 4 | 3 | 6 | 6
Participants
  Partial Response | 0 | 0 | 1 | 1 | 0 | 0
  Partial Response Unconfirmed | 0 | 0 | 0 | 0 | 1 | 0
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 28-days per cycle up to 9 months plus a 30-day follow-up period for a total of approximately up to 10 months.
Description: Analysis population consists of all participants who received at least one dose of study treatment.
Arm/Group | MK-8353 100 mg Twice Daily (BID) | MK-8353 200 mg BID | MK-8353 300 mg BID | MK-8353 350 mg BID | MK-8353 400 mg BID | MK-8353 800 mg BID
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/3 | 1/4 | 0/3 | 1/7 | 2/6
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/3 | 1/4 | 1/3 | 3/7 | 5/6
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 4/4 | 3/3 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8353 100 mg Twice Daily (BID) (N=2) | MK-8353 200 mg BID (N=3) | MK-8353 300 mg BID (N=4) | MK-8353 350 mg BID (N=3) | MK-8353 400 mg BID (N=7) | MK-8353 800 mg BID (N=6)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8353 100 mg Twice Daily (BID) (N=2) | MK-8353 200 mg BID (N=3) | MK-8353 300 mg BID (N=4) | MK-8353 350 mg BID (N=3) | MK-8353 400 mg BID (N=7) | MK-8353 800 mg BID (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VITREOUS FLOATERS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 3 (4) | 2 (3) | 4 (4)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERUCTATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 3 (3)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
FACE OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (5) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
BLOOD ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD BILIRUBIN (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (3) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATININE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATININE ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
AMNESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (9) | 2 (2) | 3 (6) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication, presentation, or any media that report any results of the trial.